CLINICAL TRIAL: NCT03997565
Title: Motor Performance Modulation After Total Knee Replacement
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 749
Record Dates: First submitted 2019-06-10; First posted 2019-06-25 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Total Knee Replacement

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients TKR
  Interventions: Procedure: TKR
- Healthy subjects

INTERVENTIONS:
Procedure: TKR — No intervention provided, but investigation of the ability to modulate motor performance during specific and functional tasks in subjects undergoing TKR compared with healthy subjects.
  Groups: Patients TKR

SUMMARY:
Functional recovery after total knee replacement (TKR) is characterized by an incomplete muscle strength due to arthrogenic muscle inhibition (AMI) and tendency to estimate the functional level. These deficits could be related to alteration of sensory feedback, and could influence the ability to modulate patients' motor performance.

To date, there are not studies investigatin the ability to modulate the motor performance in patients with TKR compared to healthy age-matched subjects.

In this study 20 patients with TKR and 20 healthy will be included . Inclusion criteria are: age between 40 and 80 , TKR for primary knee osteoarthritis, knee flexion ≥ 90° and complete knee extension, ability to perform a sit to stand on a 46 cm high chair and to walk for at least 50 meters without aids. Exclusion criteria: patients undergoing TKR after traumas, previous tibial or femoral osteotomy, partial or complete revision surgery. subjects with psychiatric and/or cognitive impairments, or with neurological, musculoskeletal or other disorders that could influence motor or functional recovery will be also exluded.

The aim of the study is to investigate the ability in motor performance modulation in patients after TKR compared to healthy age-mtched subjects.

Primary endpoint is to investigate this ability during a leg extension performed in open kinetic chain. This ability will be also evaluated during a Sit To Stand and during walking (with 10 Meters Walking Test). Secondary endpoint is to investigate pain, rate of perceived exertion and perceived load symmetry during the three tests. In both healthy and TKR groups these outcomes will be detected two times. In particular, in TKR group, patients will be tested the day before surgery and 5 days after surgery.

This study is aimed at conducting a survey in healthy subjects and in a population of subjects undergoing TKR . Participants will undergo an acquisition similar to others already described in the literature and without adverse events. Tests will last about 60 minutes and during them, will be used the equipment of Motion Analysis Lab of "Humanitas Research Hospital".

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 80 years
* TKR because of primary gonarthrosis
* Flexion ≥ 90° and complete knee extension
* Able to perform a Sit to Stand from a 46 cm high chair, without upper limb use
* Able to walk at least 50 meters without walking aids

Exclusion Criteria:

* TKR because of traumatic event
* Patients undergone to tibial or femoral osteotomy
* Partial or Total TKR revision
* Cognitive and psychiatric impairments
* Presence of neurological, internist or musculoskeletal system pathologies that may affect functional or motor recovery

Healthy subjects will have to comply with all the eligibility criteria just mentioned except for the inclusion criterion: Intervention of TKR following primary gonarthrosis

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients: subjects undergoing total knee replacement intervention because of primary gonarthrosis.
  Healty subjects: people with no known significant health problems who are recruited to participate as controls for a patient Group.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Change in Peak Torque (PT) in N*m | Patients will be evaluated the day before (T0) and the fifth day after surgery (T1), whereas healthy subjects will perform two evaluations, the first one at T0 and the second one 5 days after (T1)
  Force reproduction error between the PT-target and the PT-observed during knee extension with an isokinetic dynamometer (Ω = 60 °/s)

SECONDARY OUTCOMES:
Change in Overshoot (OS) in N | Patients will be evaluated the day before (T0) and the fifth day after surgery (T1), whereas healthy subjects will perform two evaluations, the first one at T0 and the second one 5 days after (T1)
  The error between OS-target and OS-observed during Sit-to-Stand using two force platforms.
Change in Walking speed (WS) in m/s | Patients will be evaluated the day before (T0) and the fifth day after surgery (T1), whereas healthy subjects will perform two evaluations, the first one at T0 and the second one 5 days after (T1)
  Error between "target speed" and "observed speed" during 10 meters walking test
Change in pain using Visual Analogue Scale (VAS) | Patients will be evaluated the day before (T0) and the fifth day after surgery (T1), whereas healthy subjects will perform two evaluations, the first one at T0 and the second one 5 days after (T1)
  Pain will be assessed with Visual Analogue Scale (VAS 0-10) ranging from 0 (absence of pain) to 10 (maximum pain)
Change in exertion using Modified Borg Scale | Patients will be evaluated the day before (T0) and the fifth day after surgery (T1), whereas healthy subjects will perform two evaluations, the first one at T0 and the second one 5 days after (T1)
  Perceived exertion will be assessed with Modified Borg Scale (0-10), ranging from 0 (no exertion) to 10 (maximum exertion)
Change in perceived body weight distribution using Visual Analogue Scale (VAS) | Patients will be evaluated the day before (T0) and the fifth day after surgery (T1), whereas healthy subjects will perform two evaluations, the first one at T0 and the second one 5 days after (T1)
  Perceived symmetry of load will be assessed with Visual Analogue Scale (VAS), ranging from -10 (body weight on left limb) to 10 (body weight on right limb). A value of 0 denotes perfect symmetry.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milano, Italy

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-07): https://cdn.clinicaltrials.gov/large-docs/65/NCT03997565/Prot_SAP_000.pdf